CLINICAL TRIAL: NCT03917394
Title: Efficacy and Safety of Erythropoietin And/Or Intravenous Iron Sucrose For Treatment of Anemia In Hip and Knee Arthroplasty: A Single-center Retrospective Study
Brief Title: Erythropoietin And/Or Iron Sucrose For Perioperative Anemia Management In Hip and Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wei Wang, MD & PhD, Clinical Professor, Peking Union Medical College Hospital
Other Study IDs: EPO-retro-cohort-PUMCH
Record Dates: First submitted 2019-04-04; First posted 2019-04-17 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Anemia, Iron Deficiency
Keywords: THA/TKA; Perioperative anemia; rHuEPO; iron sucrose
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferric Oxide, Saccharated; ferryl iron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- rHuEPO monotherapy group: rHuEPO was administrated during hospitalization period.
  Interventions: Drug: rHuEPO
- iron sucrose monotherapy group: Iron sucrose was administrated during hospitalization period.
  Interventions: Drug: Iron sucrose
- rHuEPO combined with iron sucrose group: rHuEPO combined with iron sucrose was administrated during hospitalization period.
  Interventions: Drug: rHuEPO; Drug: Iron sucrose
- control group: Subjects didn't be administrated with rHuEPO and/or iron sucrose during hospitalization period.

INTERVENTIONS:
Drug: rHuEPO — rHuEPO was administrated daily with 10000 IU or 20000 IU
  Other Names: Recombinant Human Erythropoietin Injection
  Groups: rHuEPO combined with iron sucrose group; rHuEPO monotherapy group
Drug: Iron sucrose — Iron sucrose was administrated daily with 100mg or 200mg
  Other Names: IV iron
  Groups: iron sucrose monotherapy group; rHuEPO combined with iron sucrose group

SUMMARY:
Perioperative anemia is very common in patients undergoing total hip arthroplasty (THA) and total knee arthroplasty (TKA). This study retrospectively analyzes the use of rHuEPO and iron sucrose in patients undergoing total hip and knee arthroplasty in order to observe the short-term efficacy and safety of rHuEPO and iron sucrose.

DETAILED DESCRIPTION:
This study aims to explore whether short-term use of rHuEPO and iron sucrose can improve postoperative anemia and promote postoperative rehabilitation after hip and knee arthroplasty. According to different therapies of perioperative anemia , included subjects would be divided into rHuEPO monotherapy group, iron sucrose monotherapy group, rHuEPO combined with iron sucrose group and control group (without rHuEPO and iron sucrose).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent hip or knee arthroplasty between May 1, 2012 (included) and December 31, 2015 in Peking Union Medical College Hospital
2. Age ≥ 18 years, sex unlimited

Exclusion Criteria:

1. Patients with serious absence of clinical data
2. Patients with rHuEPO contraindication

   1. Patients with uncontrolled severe hypertension
   2. Patients allergic to this product and other mammalian cell derivatives, or to human serum albumin
   3. Co-infected patients
3. Patients definitely allergic to iron sucrose injection
4. Patients with coagulation dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total hip and knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 780 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Differences in changes of Hb level in rHuEPO, iron sucrose, rHuEPO combined with iron sucrose and control group. | Operation day to postoperative day 7
  Changes of Hb level =Hb level in postoperative 7d - Hb level in operation day

SECONDARY OUTCOMES:
Differences in change of red blood cells count(RBC) in rHuEPO, iron sucrose, rHuEPO combined with iron sucrose and control group. | Operation day to postoperative day 7
  Changes of RBC =RBC in postoperative day 7 - RBC in operation day
Differences in change of hematokrit (HCT) in rHuEPO, iron sucrose, rHuEPO combined with iron sucrose and control group. | Operation day to postoperative day 7
  Changes of HCT =HCT level in postoperative day 7 - HCT level in operation day
Differences in change of allogeneic transfusion rate(%) in rHuEPO, iron sucrose, rHuEPO combined with iron sucrose and control group. | Operation day to postoperative day 7
  Transfusion rate is defined as the ratio of numbers subjected to blood transfusion in each group subjects.
  Blood transfusion volume is defined as the amount of blood transfusion during operation day and postoperative period.
Differences in change of allogeneic blood transfusion volume in rHuEPO, iron sucrose, rHuEPO combined with iron sucrose and control group. | Operation day to postoperative day 7
  Allogeneic blood transfusion volume is defined as the amount of blood transfusion volume from operation day to postoperative day 7 Blood transfusion volume is defined as the amount of blood transfusion during operation day and postoperative period.
Difference in postoperative hospital days in rHuEPO, iron sucrose, rHuEPO combined with iron sucrose and control group. | Up to 4 months
  Postoperative hospital days is defined as the number of days from operation day to hospital discharge.
Comparing differences of blood loss volume in each group. | Operation day to postoperative day 7
  Blood loss volume is defined as the total volume of intraoperative bleeding and postoperative drainage.
Comparing the rate of anemia between operation day and post-operation day 7 in each group. | Operation day to postoperation day 7
  According to 2011 World Health Organization(WHO) anemia standard，Hb< 130g/L for adult men and Hb < 120g/L for non-pregnant women are defined as anemia.
Differences in changes of platelet count in rHuEPO, iron sucrose, rHuEPO combined with iron sucrose and control group. | Operation day to postoperative day 7
  Changes of platelet count =platelet count in postoperative 7d - platelet count in operation day
Safety of rHuEPO and/or iron sucrose | Form operation day to postoperative day 7
  Adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watts CD, Pagnano MW. Minimising blood loss and transfusion in contemporary hip and knee arthroplasty. J Bone Joint Surg Br. 2012 Nov;94(11 Suppl A):8-10. doi: 10.1302/0301-620X.94B11.30618. PMID 23118371
- [Background] Na HS, Shin SY, Hwang JY, Jeon YT, Kim CS, Do SH. Effects of intravenous iron combined with low-dose recombinant human erythropoietin on transfusion requirements in iron-deficient patients undergoing bilateral total knee replacement arthroplasty. Transfusion. 2011 Jan;51(1):118-24. doi: 10.1111/j.1537-2995.2010.02783.x. PMID 20624257
- [Background] Conlon NP, Bale EP, Herbison GP, McCarroll M. Postoperative anemia and quality of life after primary hip arthroplasty in patients over 65 years old. Anesth Analg. 2008 Apr;106(4):1056-61, table of contents. doi: 10.1213/ane.0b013e318164f114. PMID 18349173
- [Background] Bou Monsef J, Boettner F. Blood management may have an impact on length of stay after total hip arthroplasty. HSS J. 2014 Jul;10(2):124-30. doi: 10.1007/s11420-014-9384-x. Epub 2014 Apr 8. PMID 25050095
- [Background] Lin DM, Lin ES, Tran MH. Efficacy and safety of erythropoietin and intravenous iron in perioperative blood management: a systematic review. Transfus Med Rev. 2013 Oct;27(4):221-34. doi: 10.1016/j.tmrv.2013.09.001. Epub 2013 Oct 15. PMID 24135037
- [Background] Voorn VM, van der Hout A, So-Osman C, Vliet Vlieland TP, Nelissen RG, van den Akker-van Marle ME, Dahan A, Marang-van de Mheen PJ, van Bodegom-Vos L. Erythropoietin to reduce allogeneic red blood cell transfusion in patients undergoing total hip or knee arthroplasty. Vox Sang. 2016 Oct;111(3):219-225. doi: 10.1111/vox.12412. Epub 2016 Jun 17. PMID 27314459
- [Background] Tran DH, Wong GT, Chee YE, Irwin MG. Effectiveness and safety of erythropoiesis-stimulating agent use in the perioperative period. Expert Opin Biol Ther. 2014 Jan;14(1):51-61. doi: 10.1517/14712598.2014.858116. Epub 2013 Nov 13. PMID 24219367
- [Background] Li Y, Yin P, Lv H, Meng Y, Zhang L, Tang P. A meta-analysis and systematic review evaluating the use of erythropoietin in total hip and knee arthroplasty. Ther Clin Risk Manag. 2018 Jul 10;14:1191-1204. doi: 10.2147/TCRM.S159134. eCollection 2018. PMID 30022832
- [Background] Crosby E. Perioperative use of erythropoietin. Am J Ther. 2002 Sep-Oct;9(5):371-6. doi: 10.1097/00045391-200209000-00003. PMID 12237728
- [Background] Clevenger B, Richards T. Pre-operative anaemia. Anaesthesia. 2015 Jan;70 Suppl 1:20-8, e6-8. doi: 10.1111/anae.12918. PMID 25440391
- [Background] Munoz M, Acheson AG, Auerbach M, Besser M, Habler O, Kehlet H, Liumbruno GM, Lasocki S, Meybohm P, Rao Baikady R, Richards T, Shander A, So-Osman C, Spahn DR, Klein AA. International consensus statement on the peri-operative management of anaemia and iron deficiency. Anaesthesia. 2017 Feb;72(2):233-247. doi: 10.1111/anae.13773. Epub 2016 Dec 20. PMID 27996086
- [Background] Munoz M, Gomez-Ramirez S, Cuenca J, Garcia-Erce JA, Iglesias-Aparicio D, Haman-Alcober S, Ariza D, Naveira E. Very-short-term perioperative intravenous iron administration and postoperative outcome in major orthopedic surgery: a pooled analysis of observational data from 2547 patients. Transfusion. 2014 Feb;54(2):289-99. doi: 10.1111/trf.12195. Epub 2013 Apr 15. PMID 23581484